CLINICAL TRIAL: NCT02835729
Title: A Phase 1 Trial of Indoximod in Combination With Idarubicin and Cytarabine in Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: A Study of Indoximod in Combination With (7+3) Chemotherapy in Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLG2106
Record Dates: First submitted 2016-07-11; First posted 2016-07-18 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1a (Experimental): Patients enrolled in this arm will receive standard induction and consolidation chemotherapy (7+3) with Indoximod (freebase formulation). These patients will additionally receive maintenance therapy with indoximod for 6 months after consolidation therapy. The indoximod dose will be studied in up to 4 dose levels.
  All current subjects will transition from indoximod freebase capsules over to indoximod HCL F2 tablets. All new subjects enrolled will also receive indoximod HCL F2 tablets.
  Interventions: Drug: Idarubicin; Drug: Cytarabine; Drug: Indoximod Freebase; Drug: Indoximod HCL F2
- Phase 1b (CLOSED TO ACCRUAL) (Experimental): Patients enrolled in this arm will receive standard induction and consolidation chemotherapy (7+3) with Indoximod (HCL F1 formulation). These patients will receive maintenance therapy with indoximod for 6 months after consolidation therapy. The indoximod dose will be studied in up to 4 dose levels.
  Interventions: Drug: Idarubicin; Drug: Cytarabine; Drug: Indoximod HCL F1

INTERVENTIONS:
Drug: Idarubicin — Chemotherapy
Drug: Cytarabine — Chemotherapy
Drug: Indoximod Freebase — IDO pathway inhibitor
  Arms: Phase 1a
Drug: Indoximod HCL F1 — IDO pathway inhibitor
  Arms: Phase 1b (CLOSED TO ACCRUAL)
Drug: Indoximod HCL F2 — IDO pathway inhibitor
  Arms: Phase 1a

SUMMARY:
The purpose of this study is to characterize the regimen limiting toxicities (RLT) and recommended Phase 2 dose (RP2D) of indoximod in patients with newly diagnosed AML receiving remission induction chemotherapy with cytarabine and idarubicin.

ELIGIBILITY:
Inclusion Criteria:

* A histologically or pathologically confirmed diagnosis of AML based on WHO classification with or without extramedullary disease except for central nervous system disease.
* ECOG performance status ≤ 2
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Female patients of childbearing potential must have a negative pregnancy test < 1 week prior to enrollment.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients receiving any other investigational agents or immunotherapy
* Patients who have received prior chemotherapy for AML with the exception of hydroxyurea or leukapheresis for leukocytosis; prior hypomethylating or immunomodulatory agents for MDS are allowed
* Previous allo-HSCT of any kind
* Active, uncontrolled infection including known hepatitis B or C
* Active autoimmune disease and chronic inflammatory conditions requiring concurrent use of any systemic immunosuppressants or steroids.
* History of any other active cancer diagnosis
* Pregnant women
* Known HIV-infected patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-07; Primary Completion 2019-10-25 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Safety assessed by development of RLT, AEs and laboratory parameters of indoximod. | 6 months
  Phase 1
Comparison of serum concentrations (Cmax/Steady State) of indoximod freebase and indoximod salt formulation. | 6 months
  Phase 1

SECONDARY OUTCOMES:
Measurable Residual Disease Rate | 2 years
Clinical response rate | 2 years
Duration of complete response | 2 years
Event free survival | 2 years
  Time on study to induction failure, relapse or death
Cumulative incidence of relapse (CIR) | 2 years
Overall survival (OS) | 2 years
Proportion of AML patients who become eligible for bone marrow transplantation | 2 years
Frequency and severity of adverse events | 2 years
Pharmacokinetics: Serum concentrations (Cmax/Steady State) | 6 months
  Characterize the pharmacokinetics (PK) of indoximod, idarubicin and cytarabine through analysis of blood samples

OTHER OUTCOMES:
Serum kynurenine and tryptophan levels | 2 years
  Characterize the pharmacodynamic (PD) effect of indoximod
IDO expression by immunohistochemistry in diagnostic and follow-up bone marrow biopsy specimens | 2 years
IDO protein and mRNA expression in diagnostic and follow-up bone marrow aspirate samples | 2 years
Methylation status of the IDO promoter in diagnostic and follow up bone marrow aspiration samples | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Augusta University, Augusta, Georgia
  - University of Maryland, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No